CLINICAL TRIAL: NCT00596245
Title: Open-Label, Placebo-Controlled, Parallel Group Study in Healthy Volunteers to Evaluate the Effects of Two Single MT 400 or Naproxen Sodium Tablets Administered Two Hours Apart on Chromosomal Aberrations in Peripheral Blood Lymphocytes
Brief Title: Open-Label, Placebo-Controlled, Parallel Group Study in Healthy Volunteers to Evaluate the Effects of Two Single MT 400 or Naproxen Sodium Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: POZEN (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MT400-108
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: non-smoking healthy volunteers aged 18 - 35

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): MT 400, naproxen sodium 550mg
  Interventions: Drug: MT400

INTERVENTIONS:
Drug: MT400 — MT 400, naproxen sodium 550mg

SUMMARY:
This is an open-label, parallel group, single-center study. The study design consists of a screening and a treatment period. A total of 42 (approximately 21 of each sex) non-smoking healthy volunteers aged 18 - 35.

DETAILED DESCRIPTION:
This is an open-label, parallel group, single-center study. The study design consists of a screening and a treatment period. A total of 42 (approximately 21 of each sex) non-smoking healthy volunteers aged 18 - 35, will be selected for treatment. Potential subjects will be assessed for exposure to ionizing radiation or working with cytotoxic chemicals, or who have cell cycle times that fall outside the range of 13 ± 1.5 hours or subjects with stable chromosomal rearrangements and/or abnormally high background chromosomal aberration frequencies. Approximately 30 subjects (10 per arm) are estimated to be needed for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are 18-35 years of age at the screening visit
2. Female subjects are eligible for participation in the study if they are of:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
   2. Childbearing potential, have a negative pregnancy test (urine) at Screening, and at least one of the following applies or is agreed to by the subject:

      * Female sterilization or sterilization of male partner; or,
      * Any non-medicated intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year; or,
      * Barrier method
3. Physical status within normal limits for age and consistent with observations at Screening
4. Subject agrees to remain sequestered on site during the treatment phase of the study and is willing and able to abstain from the consumption or use of any alcohol, caffeine containing beverages or medication for the duration of the study
5. Subject is able to understand and comply with study procedures required and able and willing to provide written informed consent prior to any study procedures being performed

Exclusion Criteria:

1. History of hypersensitivity, allergy, intolerance or contraindication to the use of any triptan, NSAID or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps and asthma
2. History or presence of cardio-or cerebrovascular disease; e.g., diabetes, hypertension, hyperlipidemia
3. History or presence of congenital heart disease, cardiac arrhythmias requiring medication, or a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in the study
4. History or evidence of any ischemic vascular diseases including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome, or sign/symptoms consistent with any of the above
5. History or evidence of central nervous system pathology including stroke and/or transient ischemic attacks, epilepsy or structural brain lesions which lower the convulsive threshold, or has been treated with an antiepileptic drug for seizure control within 5 years prior to screening
6. History or evidence of impaired hepatic or renal function or any screening laboratory assessment that is clinically significant in the investigator's opinion
7. Has clinically significant allergic disease (excluding non-active hay fever) or a history of multiple drug allergies
8. Evidence of macrocytic or microcytic anemia or deficiency of folate or B12 at Screening
9. Blood donation in excess of: 500 mL in 14 days; 1,500 mL in 180 days or 2,500 mL in one year
10. History of any bleeding disorder
11. Gastrointestinal disorder, surgery, ulceration, or perforation in the past 6 months; gastrointestinal bleeding in the past year; or evidence or history of inflammatory bowel disease
12. Females actively trying to become pregnant or breast feeding
13. History or evidence of alcohol abuse (more than 28 units of alcohol (male) or 21 units of alcohol (female) per week) or substance abuse within the last year or any concurrent medical or psychiatric condition which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicate participation in this clinical trial
14. Participated in a investigational drug trial within the previous four weeks
15. Used tobacco products within the past year
16. Has taken any medication, including over-the counter, prescription, herbal remedies, within one month of the first dose (with the exception of vitamin/mineral supplements)
17. Is currently working or living in an environment that exposes subject to cytotoxic chemicals or ionizing radiation, or subject has had any medical X-Ray, vaccination, or significant viral or bacterial illness within one month of Screening
18. Body Mass Index outside the range of 19-32 kg/m2 at Screening
19. Presence or history of any malignancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the impact on production of chromosomal aberration after dosage of MT 400 or naproxen sodium versus placebo. Comparison of post-dose chromosomal aberration rates will also be made to baseline rates within each arm. | 7 days

SECONDARY OUTCOMES:
Potential subjects will be assessed for exposure to ionizing radiation or working with cytotoxic chemicals. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Medlock, MD, Principal Investigator — PPD Development, LP
Locations (1):
- Matthew M. Medlock, MD, Austin, Texas, United States